CLINICAL TRIAL: NCT06140914
Title: Biological Mechanisms Behind Resynchronization Therapy in Heart Failure
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Marcus Stahlberg, Associate professor, MD, Region Stockholm
Other Study IDs: CRT K 2022-8295
Record Dates: First submitted 2023-11-14; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure; Cardiac Remodeling, Ventricular
Keywords: Proteomics; miRNA; Force-calcium study
MeSH Terms: conditions — Heart Failure; Ventricular Remodeling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples Heart biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CRT: Heart failure patients that receive a CRT
  Interventions: Diagnostic Test: Proteomics, miRNA studies and studies of blood cells from blood samples
- Control: Heart failure patients treated with medicines, without a CRT indication.
  Interventions: Diagnostic Test: Proteomics, miRNA studies and studies of blood cells from blood samples

INTERVENTIONS:
Diagnostic Test: Proteomics, miRNA studies and studies of blood cells from blood samples — This is an observational study where we follow patients and save blood samples and biopsies for analysis as described above.
  Other Names: Force-calcium study from biopsy

SUMMARY:
Heart failure is a common disease, affecting 2-3% of the population in the western world. About 30% of patients with heart failure and reduced ejection fraction display signs of electrical dyssynchrony on ECG, usually left bundle branch block (LBBB), which is associated with a worse prognosis. Cardiac resynchronization therapy (CRT) reduce mortality for patients with dyssynchronic heart failure, defined as ejection fraction (EF) = or < 35% and LBBB. About 1/3 of the patients that fit CRT criteria will not respond to CRT. Which patients that will turn out to be non-responders cannot be anticipated beforehand.

We have started a clinical study to collect blood samples, heart tissue and clinical data from heart failure patients eligible for CRT and a control group of heart failure patients on medical therapy. Patients will be assessed before CRT implantation or early after initiation of medical treatment, at 3 months, 6 months and 12 months.

Blood samples and tissue will be analysed in the search for (i) biomarkers to separate CRT responders from non-responders and (ii) mechanisms behind the remodelling observed in CRT and with medical therapy.

DETAILED DESCRIPTION:
In dyssynchrony the conduction of electrical signals within the heart is prolonged causing a delay between the activation and contraction of septum and lateral left ventricular wall. In turn, this results in uncoordinated and ineffective heart work. Dyssynchrony is accompanied by cardiac remodeling with dilatation of the left chamber. Whether dilatation is an effect or a cause of dyssynchrony is unclear and likely different for different patients. Cardiac resynchronization therapy, CRT, is a pacemaker with an extra electrode that will stimulate the right and left ventricle simultaneously, resulting in resynchronization.

We have started a clinical study to collect blood samples, heart tissue and clinical data (echocardiography, ECG, medical records) from heart failure patients eligible for CRT and a control group of heart failure patients on medical therapy. Patients will be assessed before CRT implantation or early after initiation of medical treatment, at 3 months, 6 months and 12 months. A subset of the patients in the CRT group will also also be subjected to a heart biopsy before CRT implantation and at 3 months. At each time point all patients will be assessed with echocardiography, ECG and blood sampling. The blood samples will be analyzed regarding proteins and exosomal miRNA. The heart tissue will be frozen and analyzed regarding proteins, RNA and contractility.

Endothelial function is also known to play a crucial role in heart failure and will be evaluated at inclusion, 3 and 12 months using EndoPAT. Red blood cells (RBCs) are collected to determine whether they may affect endothelial cell function.

ELIGIBILITY:
Inclusion Criteria:

1. Ejection fraction (EF) = or < 35% and A or B

   A) Left bundle branch block (LBBB) QRS = or > 150 ms or a high proportion ventricular pacing and planned for CRT at Karolinska University Hospital.

   B) Planned for medical treatment and followed at Karolinska University Hospital.
2. Ability to understand the given information.
3. Ability to give informed consent.

Exclusion Criteria:

1. Pregnant or planning pregnancy
2. Not able to give informed consent -

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Heart failure patients followed at the Karolinska University Hospital in Stockholm, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Biomarkers | 2023-2028
  Proteins or exosomal miRNA from blood to separate CRT responders from non-responders

SECONDARY OUTCOMES:
Endothelial function | 2023-2028
  EndoPAT and RBC studies to separate CRT responders from non-responders

OTHER OUTCOMES:
Mechanism behind the reverse remodelling in CRT responders and with medical treatment | 2023-2028
  Proteomics, RNA studies, force-calcium studies

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Ståhlberg, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska Universitetssjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No